CLINICAL TRIAL: NCT07250451
Title: The Effect Of Multiple Scenarios Simulation Education And Clinical Practice On Nursing Students' Competence: Quasi Experimental Crossover Study
Brief Title: Simulation Education and Clinical Practice on Nursing Students' Competence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duzce University (Other)
Responsible Party: Principal Investigator, Atiye Erbaş, Assistant Professor, Duzce University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: DU-AE-01
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Health Knowledge, Attitudes, Practice
Keywords: nursing education; Simulation practice; nursing students
MeSH Terms: conditions — Behavior | interventions — Training Support

STUDY DESIGN:
Intervention Model Description: This study used a quasi-experimental, randomized, crossover design. All groups were exposed to both simulation-based training and clinical practice in different sequences. Each student participated in both intervention conditions at different time points, allowing within-subject comparison of competence outcomes. The study used a quasi-experimental, randomized, crossover design. After obtaining written consent, students who agreed to participate were stratified by gender and randomly assigned to one of three groups (A, B, or C) by a blinded faculty member to avoid allocation bias.
  Group A: Participated in four simulation days followed by eight clinical practice days.
  Group B: Completed four clinical practice days, then four simulation days, and finally four additional clinical practice days.
  Group C: Completed eight clinical practice days followed by four simulation days.
Who Masked: Outcomes Assessor
Masking Description: This study was conducted as an open-label educational intervention. Neither participants nor researchers were blinded to group assignment due to the nature of the simulation and clinical training interventions. Data were entered into a statistical program and analyzed by an expert statistician who was blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Simulation-First Hybrid Training (Experimental): Students in Simulation-First Hybrid Training participated in four days of simulation-based training followed by eight days of clinical practice. Simulation sessions were conducted in subgroups of 4-5 students, followed by debriefing sessions. Clinical practice was conducted in hospital settings under faculty supervision.
  Interventions: Other: Educational/training
- Clinical Practice-Simulation-Clinical Practice (Integrated Training) (Experimental): Students in Clinical Practice-Simulation-Clinical Practice (Integrated Training) first completed four days of clinical practice, then four days of simulation-based training, followed by an additional four days of clinical practice. Simulation and clinical practice sessions were conducted as described for Simulation-First Hybrid Training.
  Interventions: Other: Educational/training
- Clinical Practice-First Training Followed by Simulation (Experimental): Students in Clinical Practice-First Training Followed by Simulation completed eight days of clinical practice, followed by four days of simulation-based training. Simulation and clinical practice sessions were conducted as described for Simulation-First Hybrid Training.
  Interventions: Other: Educational/training

INTERVENTIONS:
Other: Educational/training — Simulation-First Hybrid Training - Simulation → Clinical Practice:
  Students first participated in four days of simulation in subgroups of 4-5, using low-fidelity mannequins for scenarios such as colorectal surgery care, subdural hematoma, BPH surgery, coronary bypass, femur fracture, and total laryngectomy. Prebriefing and debriefing (GAS method) were conducted. This was followed by eight days of clinical practice under faculty supervision.
  Clinical Practice-Simulation-Clinical Practice (Integrated Training) - Clinical Practice → Simulation → Clinical Practice:
  Students completed four days of clinical practice, four days of simulation as above, then four additional clinical practice days.
  Clinical Practice-First Training Followed by Simulation - Clinical Practice → Simulation:
  Students completed eight days of clinical practice followed by four days of simulation. Simulation sessions and clinical practice were conducted under faculty supervision.

SUMMARY:
The aim of this study is to determine the effect of integrated education, combining clinical practice and simulation laboratory training, on the competence of second-year undergraduate nursing students. This research is designed as a multi-crossover quasi-experimental randomized controlled study. In this model, all groups were exposed to simulation training sessions in specific stages. This design is currently used in the clinical practice component of the Surgical Nursing course. Additionally, the researchers aimed to answer the question: "What is the most appropriate timing for simulation training to enhance nursing students' competence?"

During the clinical practice of the Surgical Diseases Nursing course, approximately 29-33 students participated in the simulation laboratory sessions, while about 61-65 students were involved in clinical field practice. For the simulation sessions, subgroups consisting of 4-5 students were formed. After each subgroup completed the simulation practice, a debriefing session was conducted. Each simulation scenario and related training lasted approximately half a day.

DETAILED DESCRIPTION:
This study aims to evaluate the effect of integrating simulation-based laboratory sessions with clinical practice on the competence of second-year undergraduate nursing students enrolled in the Surgical Nursing course. The study was designed as a quasi-experimental, randomized, multi-crossover study model. In this design, all student groups were sequentially exposed to simulation-based training integrated within the clinical education process, allowing each group to experience both simulation and clinical practice in different sequences.

Setting

The laboratory environment was located on the first floor of the Faculty of Health Sciences. It was arranged as a patient room and equipped with two full-body low-fidelity mannequins and all necessary nursing materials for patient care. The lab had a capacity of 15-17 students and included a separate area with chairs and a whiteboard for debriefing and discussion sessions. Before each simulation, the environment and mannequins were prepared in accordance with the specific scenario. Simulation implementation and debriefing were conducted by the first author, while clinical practice supervision was carried out by the other three researchers.

Simulation Scenarios

A total of seven different low-fidelity simulation scenarios were used, including:

Preoperative preparation and postoperative care in colorectal surgery,

Postoperative care after subdural hematoma surgery,

Postoperative care after benign prostatic hyperplasia surgery,

Postoperative care after coronary bypass surgery,

Care of a patient with femur fracture,

Postoperative care after total laryngectomy.

All scenarios were developed based on the literature and reviewed by experts for content validity. Pilot testing was conducted during the previous academic year, and minor revisions were made based on feedback.

Briefing and Prebriefing

One week before each simulation, the theoretical content related to the upcoming scenario was taught to all students using traditional classroom instruction, and relevant course materials were provided. Students scheduled for the next simulation were informed of their specific scenario in advance and were asked to review the materials again. Prior to the simulation, the laboratory environment was introduced, and students were given 5-10 minutes to familiarize themselves with the setting. They were also informed that they could withdraw from the activity if they felt psychologically uncomfortable at any time.

Simulation Implementation

Students participated in groups of 4-5. Each group entered the lab as if entering a real patient room, greeted the patient (represented by the mannequin), and provided nursing care based on the patient's vital signs, lab results, and clinical complaints. In some scenarios, such as femur fracture care, complications like fat embolism were introduced to enhance realism. Students were expected to respond to these acute situations in addition to performing routine care. Each simulation lasted approximately 20-25 minutes. At the end of each scenario, students conducted patient handover to the next group (shift), ensuring continuity of care similar to real clinical practice. The patient's voice was provided by the first researcher.

Debriefing

Following each simulation, all four subgroups were brought together for a structured debriefing session based on the Gather-Analyze-Summarize (GAS) model. This session was designed to facilitate reflection, discussion of decision-making processes, and consolidation of learning outcomes.

Data were collected before and after the interventions using validated nursing competence measurement tools. The findings are expected to contribute to the optimization of simulation-based learning strategies in nursing education and to provide evidence for the effective timing and integration of simulation training within clinical education.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate nursing students enrolled in the second year of the program
* Willing to participate in the study

Exclusion Criteria:

* Students under 18 years of age
* Students who do not provide voluntary consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Nursing Competence | up to 12 weeks
  The primary outcome is the level of nursing competence of second-year undergraduate nursing students, measured using a validated Nursing Competence Scale. Competence assessment includes clinical skills, decision-making, and ability to apply theoretical knowledge in simulation and clinical practice settings.
Simulation Learning | up to 12 weeks
  Learning outcomes specific to simulation sessions were assessed using the Simulation Learning Evaluation Scale. This scale measures students' understanding, performance, and ability to apply skills in the simulated environment. Administered to each laboratory subgroup after simulation.

SECONDARY OUTCOMES:
Demographic Data | Baseline (pre-intervention)
  Demographic information including age, gender, and academic background was collected from all participants using a structured demographic form before clinical practice.

CONTACTS AND LOCATIONS:
Locations (1):
- Duzce University, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
ndividual participant data will not be shared due to privacy and ethical considerations of student participation.